CLINICAL TRIAL: NCT04815668
Title: Effect of Acupuncture at the Sphenopalatine Ganglion in the Treatment of Moderate-to-severe Seasonal Allergic Rhinitis
Brief Title: Acupuncture at the Sphenopalatine Ganglion in the Treatment of Moderate-to-severe Seasonal Allergic Rhinitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Aerospace 731 Hospital (Other)
Responsible Party: Principal Investigator, weiming wang, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020YK14
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Intervention Model Description: Participants who agreed to randomization will be allocated to the acupuncture group, sham acupuncture group or rescue medication group in a 1:1:1 ratio
Who Masked: Investigator, Outcomes Assessor
Masking Description: the participants in acupuncture group and SA group, outcome evaluators and statistician in the two acupuncture groups will be blinded to the group allocation throughout the entire trial. Participants in the rescue medication group and acupuncturists will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture group (Experimental)
  Interventions: Other: Acupuncture group
- Placebo acupuncture group (Placebo Comparator)
  Interventions: Other: Placebo acupuncture group
- Rescue medication (Other)
  Interventions: Other: Rescue medication group

INTERVENTIONS:
Other: Acupuncture group — Sterile single-use stainless steel needles (size 0.35 mm × 55 mm) (YiDaiFu brand, Suzhou Tianyi Acupuncture Instrument Co., Ltd., Suzhou, China) will be utilized. Participants in lateral position, the acupoints area will be sterilized with 75% alcohol. To stimulate SPG, the needles will be inserted in the medial superior anterior direction to a depth of approximately 55 mm33 until the participants report a special sensation radiating toward the nose or the upper teeth. After that, the needle will be withdrew slightly. The needles will be retained for 30 minutes after three stimulation. Rescue medication are permitted when participants feel that their symptoms are intolerable.
  Arms: Acupuncture group
Other: Placebo acupuncture group — The acupuncture procedure will be similar to that of the acupuncture group. After sterilizing the skin, the 0.35 × 25 mm disposable needle will be vertically inserted at SPG acupoint about 3-5 mm. No needle manipulation will be conducted to avoid the deqi response. Rescue medication are permitted when participants feel that their symptoms are intolerable.
  Arms: Placebo acupuncture group
Other: Rescue medication group — Participants in the rescue medication group do not receive acupuncture treatment during the study period. They will be only allowed to use rescue medication. They have the option of 4 weeks (up to 8 sessions) of acupuncture free of charge at the end of the follow-up period.
  Arms: Rescue medication

SUMMARY:
Allergic rhinitis (AR) is an immunoglobulin E-mediated inflammatory disease1 caused by hypersensitivity of the immune system to an allergen, affecting 100 million people in Europe 2and 400 million of the global population.The etiology of AR is multifactorial, resulting primarily from genetic predisposition, immunological response, and environmental pollutants.AR traditionally has been classified as seasonal (SAR) or perennial (PAR) depending on the causes and duration of symptoms. Some patients with AR prefer complementary and alternative medicine for their symptoms, with nearly 20% receiving acupuncture. According to the updated practice parameter of rhinitis in 2020, the use of acupuncture for the treatment of AR was not recommended due to a lack of well-controlled studies.

The sphenopalatine ganglion (SPG), located under a thin (1-2 mm) layer of mucosa in the pterygopalatine fossa, consists of sensory fibers that innervate the nasopharynx, nasal cavity, and palate.Several studies have reported the benefit of SPG stimulation in chronic cluster headache and acute ischaemic stroke. Compared with traditional acupoints selected on basis of traditional meridian theory, acupuncture at SPG(inserting a needle through SPG acupoint (near ST7, Xiaguan) to reach and directly stimulate the SPG) may help patients ameliorate nasal symptoms immediately and improve quality of life by increasing sympathetic nerve excitability, but the evidence is inconclusive.

We have designed this three-armed, randomized trial to investigate the efficacy and safety of acupuncture at SPG for the treatment of SAR. We hypothesize that acupuncture at SPG plus rescue medication is superior to sham acupuncture plus RM and RM alone in the treatment of SAR.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤ 75 years;
2. History of moderate to severe SAR symptoms (Visual analog scale(VAS) >50 mm, range, 0 cm[not at all bothersome] to 100 mm[extremely bothersome]) for more than 4 days/weeks, and more than 4 consecutive weeks with at least two years' duration;
3. Positive skin prick test to grass and birch pollen or/and serum-specific IgE test;
4. Ability to complete the medical information form and sign a written informed consent.

Exclusion Criteria:

1. History or current evidence of perennial allergic rhinitis, acute sinusitis, allergic asthma, pneumonia; autoimmune disorders, or severe chronic inflammatory diseases;
2. History of nasal rhinopolypus or abnormalities;
3. Intake of antihistamines, anticholinergics, corticosteroids, decongestants, or antibiotics during the 1 month prior to beginning the study;
4. History of systemically administered corticosteroids within 6 months or specific immunotherapy, allergy desensitization therapy within 1 year before enrollment;
5. Serious uncontrolled blood coagulation disorder, cardiovascular disorder, severe hepatic/renal insufficiency or mental disorder;
6. Pregnancy or planning for pregnancy;
7. Known allergy, or contraindication to rescue medication or related drugs;
8. Known phobia to acupuncture or having received acupuncture treatment, or sphenopalatine ganglion stimulation or other complementary and alternative medicine within 1 months prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the average daily Combined Symptoms and Medication Score (CSMS) over weeks 1- 4 | weeks 1-4
  The average daily Combined Symptoms and Medication Score (CSMS) is the sum of the daily symptom score (dSS) plus daily medication score (dMS) . The dSS contains a 6-item scale referring to nasal symptoms (4 items) and ocular symptoms (2 items), with each item scored using a Likert scale of 0 to 3. The dSS will be calculated as a mean of all non-missing dSS divided by the number of individual symptoms (range, o to 3). The dMS will again be calculated as an average of daily symptom relief medication score, with a range of 0 to 3.

SECONDARY OUTCOMES:
The change from baseline in the average daily Combined Symptoms and Medication Score (CSMS) over weeks 5- 8 and the first week following symptoms onset in the second year | over weeks 5- 8 and the first week following symptoms onset in the second year
  The average daily Combined Symptoms and Medication Score (CSMS) is the sum of the daily symptom score (dSS) plus daily medication score (dMS) . The dSS contains a 6-item scale referring to nasal symptoms (4 items) and ocular symptoms (2 items), with each item scored using a Likert scale of 0 to 3. The dSS will be calculated as a mean of all non-missing dSS divided by the number of individual symptoms (range, o to 3). The dMS will again be calculated as an average of daily symptom relief medication score, with a range of 0 to 3.
Change in the average daily symptom score (dSS) and daily medication score (dMS) from baseline over weeks 1- 4, weeks 5-8 in the first year and the first week following symptoms onset in the second year. | over weeks 1- 4, weeks 5-8 in the first year and the first week following symptoms onset in the second year.
  The daily symptom score (dSS) contains a 6-item scale referring to nasal symptoms (4 items) and ocular symptoms (2 items), with each item scored using a Likert scale of 0 to 3. The dSS will be calculated as a mean of all non-missing dSS divided by the number of individual symptoms (range, o to 3). The daily medication score (dMS) will again be calculated as an average of daily symptom relief medication score, with a range of 0 to 3.
The proportion of participants with a minimum of 23% improvement in average daily Combined Symptoms and Medication Score (CSMS) from baseline over weeks 1-4, weeks 5-8 in the first year and at the first week following symptoms onset in the second year. | over weeks 1- 4, weeks 5-8 in the first year and the first week following symptoms onset in the second year.
  A difference of 23% on the average daily Combined Symptoms and Medication Score (CSMS) was chosen to demonstrate a minimum clinically important difference.
Change in the Rhinoconjunctivitis Quality of Life Questionnaires (RQLQ) total score and subscale scores from baseline to the end of weeks 4 and 8 in the first year and the first week following symptoms onset in the second year. | At the end of weeks 4 and 8 in the first year and the first week following symptoms onset in the second year
  The RQLQ is a well-established and validated questionnaire consisted of 28 questions covering 7 domains: sleep (3 items), practical problems (3 items), non-nasal and eye symptoms (7 items), nasal symptoms (4 items), eye symptoms (4 items), activities that have been limited by nose or eye symptoms (3 items), and emotional function (4 items). Each item will be evaluated on a 7-point rating scale ranging from 0 (no impairment) to 6 (severe impairment) during the previous week.
Change in the Visual analog scale score for the overall allergic symptoms severity from baseline to the end of weeks 4 and 8 in the first year and the first week following symptoms onset in the second year. | At the end of weeks 4 and 8 in the first year and the first week following symptoms onset in the second year
  Patients will be asked to grade the severity of allergic symptoms using the self-rated 0-100mm Visual analog scale (0, no symptoms, to 100, worst-ever symptoms, in 1-point increment).
A global evaluation in comparison to previous years by each participant at the end of weeks 4 and 8 in the first year and the first week following symptoms onset in the second year. | At the end of weeks 4 and 8 in the first year and the first week following symptoms onset in the second year
  Each participant will be asked the following question: ''Compared to your symptoms in previous grass pollen seasons, how have you felt overall in this grass pollen season? (Tick only one)". The possible answers are coded as follows：1, "Very much better"; 2, "Much better"; 3, "A little better"; 4, "No change"; 5, "A little worse"; 6, "Much worse"; and 7, "Very much worse".
Patient global evaluation of improvement at the end of weeks 4 and 8 in the first year and the first week following symptoms onset in the second year. | At the end of weeks 4 and 8 in the first year and the first week following symptoms onset in the second year
  Patient global evaluation of improvement will be rated by the participants using a 7-point Likert scale with the following options: 1, "Very much better"; 2, "Much better"; 3, "A little better"; 4, "No change"; 5, "A little worse"; 6, "Much worse"; and 7, "Very much worse" at each study visit.
The average weekly number of medication-free days during weeks 1-4, weeks 5-8 in the first year. | during weeks 1-4, weeks 5-8 in the first year
  The average weekly number of medication-free days during weeks 1-4, weeks 5-8 in the first year will be compared among three groups
The average weekly number of symptom-free days during weeks 1-4, weeks 5-8 in the first year. | during weeks 1-4, weeks 5-8 in the first year
  The average weekly number of symptom-free days during weeks 1-4, weeks 5-8 in the first year will be compared among three groups

OTHER OUTCOMES:
Participants' expectation about therapeutic benefits from acupuncture | At baseline
  Participants in the acupuncture and placebo acupuncture groups will be asked the following question: "How helpful you believe the acupuncture modality you received would be for your allergic rhinitis?"
The proportion of participants remained blinded to treatment arm in acupuncture and placebo acupuncture groups. | Five minutes after the end of the last treatment in the fourth week,
  Each participant in the acupuncture and placebo acupuncture groups will be asked the following question: "Which treatment do you think you have received (acupuncture or placebo acupuncture)?"
Incidence of adverse events | during weeks 1-8 in the first year and the first week following symptoms onset in the second year
  Any potential adverse events (AEs) will be monitored and documented in the CRFs within 24 hours after their occurrence during the treatment and follow-up period. According to their potential association with acupuncture, AEs will be categorized as acupuncture-associated AEs (e.g., subcutaneous hemorrhage, dizziness, fainting, serious pain, and local infection fainting, localized hematoma), and non-treatment-related AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Wang, MD,PhD, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- No.731 Hospital of China Aerospace Science and Industry Corporation, Beijing, China

IPD SHARING:
Plan to Share IPD: No